CLINICAL TRIAL: NCT06496984
Title: Valutazione in Ingresso Del Rischio Nutrizionale Del Paziente in SC Medicina Interna Del P.O. di Acqui Terme in Regime di Ricovero: Presa in Carico Nutrizionale Per Ottimizzare l'Outcome di Patologia Acuta e Monitoraggio Nel Post-ricovero
Brief Title: Valutazione All'Ingresso Del Rischio Nutrizionale in Pazienti Ricoverati Nel Reparto di Medicina Interna (AMIDO)
Acronym: AMIDO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Azienda Sanitaria Locale di Alessandria (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Asl22.MedI.22.02
Record Dates: First submitted 2024-06-25; First posted 2024-07-11 (Actual); Last update posted 2024-07-11 (Actual); Status verified 2024-06

CONDITIONS: Malnutrition; Hospitalized Patient
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Nutritional Intervention (Experimental): All patients with MUST 1 and 2 will be sent to the dietitian. The clinician will act on the patient's characteristics by providing different dietary therapies, such as oral nutritional supports (ONS), extra nutritional cares, diet changes without supplements and artificial nutrition.
  Interventions: Other: Nutritional intervention

INTERVENTIONS:
Other: Nutritional intervention — Diet changes with different dietary therapies, such as oral nutritional supports (ONS), extra nutritional cares, diet changes without supplements and artificial nutrition.

SUMMARY:
The aim of this study is to identify the risk of malnutrition in patients admitted to the Internal Medicine departments using the MUST screening tool. Additional aspects are to evaluate malnourished patients' characteristics and effectiveness of an early nutritional programme started during hospitalization.

DETAILED DESCRIPTION:
Malnutrition is defined as a nutritional state characterized by an excess or deficient intake of nutrients. This condition may result in a change in body composition and in organic disfunctions. Malnutrition in hospitalized patients is a condition prevalent worldwide affecting between 20% and 50% of patients at admission, with further increase expected during hospitalization. Patients hospitalized in internal medicine departments are frequently older with multimorbidity and polypharmacy, so very likely to be malnourished, but the prevalence and determinants of malnutrition remain unclear.

In AMIDO study, all patients with MUST 1 and 2 will be sent to the a dietitian. The clinician will act on the patient's characteristics by providing different dietary therapies, such as oral nutritional supports (ONS), extra nutritional cares, diet changes without supplements and artificial nutrition.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted from 1st January 2023 to 31th May 2023 at the Internal Medicine Department of the Monsignor Giovanni Galliano Hospital in Acqui Terme of the Alessandria ASL.

Exclusion Criteria:

* none

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 268 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Risk of malnutrition | Before the intervention (Baseline/T0) and at the hospital discharge, an average of 8 days after (Final/T1)
  Assessment of patients' risk of malnutrition on admission through the MUST questionnaire.

SECONDARY OUTCOMES:
Clinical conditions and malnutrition | Before the intervention (Baseline/T0) and at the hospital discharge, an average of 8 days after (Final/T1)
  Correlation between clinical outcomes of enrolled patients and level of malnutrition on admission, measured by MUST questionnaire
Gender and malnutrition | Before the intervention (Baseline/T0) and at the hospital discharge, an average of 8 days after (Final/T1)
  Correlation between gender of enrolled patients and nutritional status at the time of admission, measured by MUST questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Paola Gnerre, MD, Principal Investigator — Azienda Sanitaria Locale di Alessandria (ASL AL)
Locations (1):
- Azienda Sanitaria Locale di Alessandria (ASL AL), Alessandria, Piedmont, Italy